CLINICAL TRIAL: NCT01958827
Title: A Multicenter Open-label Study of the Human Anti-TNF Monoclonal Antibody Adalimumab to Investigate Efficacy, Safety and Pharmacokinetics After Dose Escalation in Japanese Subjects With Crohn's Disease
Brief Title: A Study of Adalimumab After Dose Escalation in Japanese Subjects With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-687; 2015-004121-13 (EudraCT Number)
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Crohn's Disease
Keywords: Dose Escalation; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab 80 mg (Experimental): All participants were to receive subcutaneous injections of open-label adalimumab 80 mg every other week from Week 0 to Week 50.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection.
  Other Names: Humira, ABT-D2E7

SUMMARY:
The purpose of this study is to investigate the efficacy, safety and pharmacokinetics after dose escalation in Japanese subjects with Crohn's Disease.

DETAILED DESCRIPTION:
Subjects who are confirmed to meet all of the inclusion criteria and none of the exclusion criteria during screening period (≤ 21 days) will be given subcutaneous injections of open-label adalimumab 80 mg eow from Week 0 to Week 50. If a subject has an inadequate response at or after Week 8, the subject may be withdrawn from the study. Self-injection of study drug is permitted for the subjects who are willing to perform self-injection, if the investigator decided as appropriate. Disease activity will be evaluated by Crohn's disease activity index (CDAI) at Screening, Week 0 and every 4 weeks until Week 52. Follow-up will be performed at 70 days after the last dose of study drug by visit or telephone.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 15 years of age at the time of informed consent.
* Subject with Crohn's disease who received induction treatment of commercially available Humira® (160 mg initially and 80 mg at 2 weeks after initial dose), achieved response after initial dose, and then lost response during maintenance treatment with Humira®.
* Subject with elevated C-reactive Protein (CRP) at Screening.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy) or is of childbearing potential and is practicing an approved method of birth control throughout the study and for 150 days after the last dose of study drug.
* Subject has a negative tuberculosis (TB) screening assessment. If the subject has evidence of a latent TB infection; the subject must initiate and complete a minimum of 21 days of an ongoing TB prophylaxis (in such case, screening period can be prolonged until 21 days past after initiation of prophylaxis and study drug is administered) or have documented completion of a full course of TB prophylaxis, prior to Week 0.

Exclusion Criteria:

* Subject with suspicion of colitis other than Crohn's disease.
* Subject with an ostomy or ileoanal pouch. (Subjects with a previous ileo-rectal anastomosis are not excluded).
* Subject with abscess or suspicion of abscess, or subject with infection(s).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morio Ozawa, MS, Study Director — AbbVie

REFERENCES:
- [Derived] Motoya S, Watanabe M, Wallace K, Lazar A, Nishimura Y, Ozawa M, Thakkar R, Robinson AM, Singh RSP, Mostafa NM, Suzuki Y, Hibi T. Efficacy and Safety of Dose Escalation to Adalimumab 80 mg Every Other Week in Japanese Patients with Crohn's Disease Who Lost Response to Maintenance Therapy. Inflamm Intest Dis. 2018 Jul;2(4):228-235. doi: 10.1159/000486786. Epub 2018 May 15. PMID 30221150
- See also: Related Info. — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 21-day screening period.
Period: Overall Study
Arm/Group | Adalimumab 80 mg
Started | 28
Completed | 18
Not Completed | 10
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 6
Not completed — Concomitant Prohibited Medicine for AE | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Response 50 (CR50; Crohn's Disease Activity Index [CDAI] Decrease ≥ 50 From Week 0) at Week 8
Description: CDAI is used to quantify the signs and symptoms of patients with Crohn's Disease. A score below 150 indicates remission and a score above 450 indicates severe disease. Non-responder imputation (NRI) for missing CDAI observations was used.
Time Frame: Week 8
Population: Full Analysis Set (FAS): All enrolled participants who received at least one dose of study drug and had at least one post-treatment efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
percentage of participants | 75 [55.1 to 89.3]

2. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (CDAI < 150) Every 4 Weeks up to Week 52
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
percentage of participants
  Week 4 | 14.3 [4.0 to 32.7]
  Week 8 | 25.0 [10.7 to 44.9]
  Week 12 | 28.6 [13.2 to 48.7]
  Week 16 | 32.1 [15.9 to 52.4]
  Week 20 | 35.7 [18.6 to 55.9]
  Week 24 | 42.9 [24.5 to 62.8]
  Week 28 | 35.7 [18.6 to 55.9]
  Week 32 | 42.9 [24.5 to 62.8]
  Week 36 | 39.3 [21.5 to 59.4]
  Week 40 | 39.3 [21.5 to 59.4]
  Week 44 | 42.9 [24.5 to 62.8]
  Week 48 | 39.3 [21.5 to 59.4]
  Week 52 | 35.7 [18.6 to 55.9]

3. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response 50 (CR50; Crohn's Disease Activity Index [CDAI] Decrease ≥ 50 From Week 0) Every 4 Weeks up to Week 52
Description: CDAI is used to quantify the signs and symptoms of patients with Crohn's Disease. A score below 150 indicates remission and a score above 450 indicates severe disease. Non-responder imputation (NRI) for missing CDAI observations was used. Week 8 was the primary outcome measure.
Time Frame: Weeks 4, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
percentage of participants
  Week 4 | 67.9 [47.6 to 84.1]
  Week 12 | 67.9 [47.6 to 84.1]
  Week 16 | 67.9 [47.6 to 84.1]
  Week 20 | 67.9 [47.6 to 84.1]
  Week 24 | 71.4 [51.3 to 86.8]
  Week 28 | 64.3 [44.1 to 81.4]
  Week 32 | 71.4 [51.3 to 86.8]
  Week 36 | 67.9 [47.6 to 84.1]
  Week 40 | 64.3 [44.1 to 81.4]
  Week 44 | 60.7 [40.6 to 78.5]
  Week 48 | 64.3 [44.1 to 81.4]
  Week 52 | 57.1 [37.2 to 75.5]

4. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response 70 (CR70; Crohn's Disease Activity Index [CDAI] Decrease ≥ 70 From Week 0) Every 4 Weeks up to Week 52
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
percentage of participants
  Week 4 | 46.4 [27.5 to 66.1]
  Week 8 | 57.1 [37.2 to 75.5]
  Week 12 | 64.3 [44.1 to 81.4]
  Week 16 | 64.3 [44.1 to 81.4]
  Week 20 | 64.3 [44.1 to 81.4]
  Week 24 | 67.9 [47.6 to 84.1]
  Week 28 | 64.3 [44.1 to 81.4]
  Week 32 | 67.9 [47.6 to 84.1]
  Week 36 | 64.3 [44.1 to 81.4]
  Week 40 | 60.7 [40.6 to 78.5]
  Week 44 | 57.1 [37.2 to 75.5]
  Week 48 | 60.7 [40.6 to 78.5]
  Week 52 | 57.1 [37.2 to 75.5]

5. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response 100 (CR100; Crohn's Disease Activity Index [CDAI] Decrease of 100 From Week 0) Every 4 Weeks up to Week 52
Description: as for outcome 1
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
percentage of participants
  Week 4 | 32.1 [15.9 to 52.4]
  Week 8 | 35.7 [18.6 to 55.9]
  Week 12 | 39.3 [21.5 to 59.4]
  Week 16 | 46.4 [27.5 to 66.1]
  Week 20 | 50.0 [30.6 to 69.4]
  Week 24 | 50.0 [30.6 to 69.4]
  Week 28 | 42.9 [24.5 to 62.8]
  Week 32 | 50.0 [30.6 to 69.4]
  Week 36 | 50.0 [30.6 to 69.4]
  Week 40 | 57.1 [37.2 to 75.5]
  Week 44 | 46.4 [27.5 to 66.1]
  Week 48 | 50.0 [30.6 to 69.4]
  Week 52 | 46.4 [27.5 to 66.1]

6. Secondary Outcome: C-reactive Protein (CRP): Mean Change From Baseline (Week 0) to Week 52
Description: C-reactive protein (CRP) was measured from blood samples as a marker for inflammation. Higher levels are indicative of more inflammation. Normal concentration in healthy human serum is usually lower than 0.3 mg/dL, slightly increasing with age. Last Observation Carried Forward (LOCF) was used for missing data.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
mg/dL
  Week 4 | -0.570 (1.4902)
  Week 8 | -0.426 (1.6072)
  Week 12 | -0.710 (1.6769)
  Week 16 | -0.923 (1.6981)
  Week 20 | -0.907 (1.7532)
  Week 24 | -0.813 (1.7924)
  Week 28 | -0.833 (1.8820)
  Week 32 | -0.853 (2.0507)
  Week 36 | -0.586 (2.3271)
  Week 40 | -1.008 (2.0471)
  Week 44 | -0.915 (2.2324)
  Week 48 | -0.649 (2.5734)
  Week 52 | -0.570 (2.7635)

7. Other Pre Specified Outcome: Change in Mean Serum Adalimumab Concentration From Baseline (Week 0) to Week 52
Description: Blood samples were drawn prior to drug administration. Adalimumab concentrations in serum were determined using a validated heterogeneous electrochemiluminescence (ECL)-immunoassay method. The assay captures adalimumab via biotinylated anti-idiotypic antibody, and detects it via sulfo-tagged TNF-alpha. n=the number of participants with available data at each time point.
Time Frame: Baseline (Week 0) to Week 52
Population: All participants in the FAS with available data at both time points.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
µg/mL
  Baseline (Week 0) (n=28) | 3.06 (2.19)
  Week 52 (n=18) | 9.47 (5.34)

8. Other Pre Specified Outcome: Change in Number of Subjects Positive for Anti-Adalimumab Antibodies (AAA) From Baseline to Week 52
Description: Serum samples with adalimumab concentration below 2 μg/mL were selected for AAA analyses. Samples were considered AAA positive if the measured AAA concentration was above 20 ng/mL. A subject was considered to be AAA positive if the subject had at least one AAA positive sample observed within 30 days following the subject's last adalimumab dose.
Time Frame: Baseline (Week 0) to Week 52
Population: FAS
Measure: Number; unit: participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
participants
  Baseline (Week 0) | 3
  Week 52 | 4

9. Secondary Outcome: Number of Participants With Potentially Significant Hematology Parameters
Description: Blood was collected for analysis at designated study visits; hematology results were provided by each site laboratory. The number of participants with an abnormal laboratory result (higher than upper limit of normal [ULN] or lower than lower limit of normal [LLN]) meeting Common Toxicity Criteria (CTC) of Grade 3 or higher is summarized. Increase is signified by ↑. n=the number of participants with CTC Grade <3 at baseline and a post-baseline value.
Time Frame: 52 weeks
Population: Safety Analysis Set: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
participants
  Haemoglobin <8 g/dL (n=27) | 1
  Haemoglobin ↑ >4.0 g/dL (n=28) | 0
  Platelet Count <5.0x10^4/mcL (n=28) | 0
  White Blood Cells <2.0x10^3/mcL (n=28) | 0
  Neutrophils <1.0x10^3/mcL(n=28) | 0
  Lymphocytes <0.5x10^3/mcL (n=28) | 4

10. Secondary Outcome: Number of Participants With Potentially Significant Clinical Chemistry Parameters
Description: Blood was collected for analysis at designated study visits; chemistry results were provided by a central laboratory. The number of participants with an abnormal laboratory result (higher than upper limit of normal [ULN] or lower than lower limit of normal [LLN]) meeting Common Toxicity Criteria (CTC) of Grade 3 or higher is summarized. n=the number of participants with CTC Grade <3 at baseline and a post-baseline value for each parameter.
Time Frame: 52 weeks
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
participants
  Alanine Aminotransferase >5xULN (n=28) | 0
  Aspartate Aminotransferase >5xULN (n=28) | 0
  Gamma-glutamyl Transpeptidase >5x ULN (n=28) | 0
  Alkaline Phosphatase >5xU/L (n=28) | 0
  Total Bilirubin >3xULN (n=28) | 0
  Creatine Phosphokinase >5x ULN (n=28) | 1
  Creatinine >3xULN or >3xBL (n=28) | 0
  Uric Acid >10.0 mg/dL (n=28) | 0
  Inorganic Phosphate <2.0 mg/dL (n=28) | 3
  Calcium <7.0 mg/dL (n=28) | 1
  Calcium >12.5 mg/dL (n=28) | 0
  Sodium <130 mEq/L (n=28) | 0
  Sodium >155 mEq/L (n=28) | 0
  Potassium <3.0 mEq/L (n=27) | 0
  Potassium >6.0 mEq/L (n=28) | 0
  Non-fasting Glucose <40 mg/dL (n=28) | 0
  Non-fasting Glucose >250 mg/dL (n=28) | 0
  Albumin <2.0 g/dL (n=28) | 0
  Cholesterol >400 mg/dL(n=28) | 0
  Triglycerides >500 mg/dL(n=28) | 0
  Magnesium <0.9 mg/dL (n=28) | 0
  Magnesium >3.0 mg/dL (n=28) | 0

11. Secondary Outcome: Systolic Blood Pressure: Mean Change From Baseline (Week 0) to Each Visit
Description: Blood pressure was measured while the participant was sitting. n=the number of participants with available data at each time point.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
mm Hg
  Week 2 (n=28) | -3.9 (11.98)
  Week 4 (n=28) | -2.5 (9.41)
  Week 8 (n=25) | -1.1 (9.98)
  Week 12 (n=21) | -1.3 (9.34)
  Week 16 (n=21) | -0.2 (11.72)
  Week 20 (n=20) | 1.9 (12.64)
  Week 24 (n=20) | 2.0 (8.89)
  Week 28 (n=20) | 0.8 (8.91)
  Week 32 (n=20) | -1.7 (7.41)
  Week 36 (n=20) | -0.5 (10.79)
  Week 40 (n=20) | 2.3 (9.55)
  Week 44 (n=19) | 1.9 (14.12)
  Week 48 (n=19) | 4.6 (11.66)
  Week 52 (n=18) | -0.3 (9.41)

12. Secondary Outcome: Diastolic Blood Pressure: Mean Change From Baseline (Week 0) to Each Visit
Description: as for outcome 11
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
mm Hg
  Week 2 (n=28) | -0.6 (9.53)
  Week 4 (n=28) | 0.2 (8.56)
  Week 8 (n=25) | 0.7 (8.13)
  Week 12 (n=21) | 1.1 (7.12)
  Week 16 (n=21) | 0.1 (7.78)
  Week 20 (n=20) | 0.8 (9.38)
  Week 24 (n=20) | 0.8 (8.72)
  Week 28 (n=20) | -0.5 (7.81)
  Week 32 (n=20) | -0.8 (9.27)
  Week 36 (n=20) | -0.4 (10.27)
  Week 40 (n=20) | 0.7 (10.66)
  Week 44 (n=19) | -1.2 (8.57)
  Week 48 (n=19) | 1.3 (8.48)
  Week 52 (n=18) | 3.0 (11.97)

13. Secondary Outcome: Heart Rate: Mean Change From Baseline (Week 0) to Each Visit
Description: Heart rate was measured while the participant was sitting. n=the number of participants with available data at each time point.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
bpm
  Week 2 (n=28) | -0.3 (11.94)
  Week 4 (n=28) | 0.7 (12.78)
  Week 8 (n=25) | -1.1 (9.48)
  Week 12 (n=21) | -1.1 (11.59)
  Week 16 (n=21) | -1.9 (9.56)
  Week 20 (n=20) | -3.0 (8.68)
  Week 24 (n=20) | -0.9 (13.15)
  Week 28 (n=20) | -1.6 (11.30)
  Week 32 (n=20) | -5.6 (11.95)
  Week 36 (n=20) | -4.7 (12.88)
  Week 40 (n=20) | -3.7 (13.88)
  Week 44 (n=19) | -2.0 (10.78)
  Week 48 (n=19) | -1.3 (15.53)
  Week 52 (n=18) | -2.8 (11.80)

14. Secondary Outcome: Body Temperature: Mean Change From Baseline (Week 0) to Each Visit
Description: n=the number of participants with available data at each time point.
Time Frame: Baseline (Week 0) and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: degrees Celcius
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
degrees Celcius
  Week 2 (n=28) | -0.03 (0.558)
  Week 4 (n=28) | -0.02 (0.571)
  Week 8 (n=25) | -0.08 (0.569)
  Week 12 (n=21) | -0.14 (0.606)
  Week 16 (n=21) | -0.11 (0.558)
  Week 20 (n=20) | -0.16 (0.545)
  Week 24 (n=20) | -0.20 (0.701)
  Week 28 (n=20) | -0.23 (0.716)
  Week 32 (n=20) | -0.26 (0.762)
  Week 36 (n=20) | -0.36 (0.476)
  Week 40 (n=20) | -0.16 (0.555)
  Week 44 (n=19) | -0.24 (0.472)
  Week 48 (n=19) | -0.03 (0.781)
  Week 52 (n=18) | -0.13 (0.717)

15. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs or TESAE) are defined as any event that began or worsened in severity after the first dose of study drug. The investigator assessed the relationship of each event to the use of study drug as either Reasonable possibility or No reasonable possibility of being related to study drug.
  For more details on adverse events please see the AE section below.
Time Frame: 60 weeks
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Adalimumab 80 mg
Number analyzed (Participants) | 28
participants
  Any TEAE | 24
  TEAEs with reasonable possibility of being related | 5
  Any severe TEAE | 2
  TESAE | 8
  Any TEAE Leading to Discontinuation of Study | 4
  Death | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of study drug administration until 70 days after last dose of study drug (60 weeks); SAEs were also collected from the time that informed consent was obtained until 70 days after last dose of study drug (up to 63 weeks).
Arm/Group | Adalimumab 80 mg
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 80 mg (N=28)
CROHN'S DISEASE (Gastrointestinal disorders) | 4
ILEUS (Gastrointestinal disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
SMALL INTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1
SUBILEUS (Gastrointestinal disorders) | 1
ANAL ABSCESS (Infections and infestations) | 1
PNEUMONIA BACTERIAL (Infections and infestations) | 1
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 80 mg (N=28)
ANAEMIA (Blood and lymphatic system disorders) | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1
CHEILITIS (Gastrointestinal disorders) | 1
DENTAL CARIES (Gastrointestinal disorders) | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
STOMATITIS (Gastrointestinal disorders) | 1
INJECTION SITE REACTION (General disorders) | 1
PYREXIA (General disorders) | 2
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
SEASONAL ALLERGY (Immune system disorders) | 1
ANAL ABSCESS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 2
CANDIDA INFECTION (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 2
MYCOPLASMA INFECTION (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 13
OTITIS EXTERNA (Infections and infestations) | 2
PERIODONTITIS (Infections and infestations) | 2
POSTOPERATIVE ABSCESS (Infections and infestations) | 1
PULPITIS DENTAL (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1
HEADACHE (Nervous system disorders) | 3
MIGRAINE (Nervous system disorders) | 1
RADICULOPATHY (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
DYSMENORRHOEA (Reproductive system and breast disorders) | 1
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 4
URTICARIA (Skin and subcutaneous tissue disorders) | 2
HYPERTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.